CLINICAL TRIAL: NCT01029353
Title: A Multi-center Randomized Trial of Laparotomy vs. Drainage as the Initial Surgical Therapy for ELBW Infants With Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP): Outcomes at 18-22 Months Adjusted Age
Brief Title: Laparotomy vs. Drainage for Infants With Necrotizing Enterocolitis
Acronym: NEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0039; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD036790 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024139 (NIH); UL1RR025744 (NIH); UL1RR025764 (NIH); UL1RR025777 (NIH); M01RR008084 (NIH); UL1RR024979 (NIH); U10HD068284 (NIH); U10HD068278 (NIH); U10HD068270 (NIH); U10HD068263 (NIH); U10HD068244 (NIH); UG1HD087226 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Enterocolitis, Necrotizing; Intestinal Perforation
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity; Laparotomy; Drainage; Isolated intestinal perforation; Focal intestinal perforation
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing; Intestinal Perforation | interventions — Laparotomy; Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Randomized Trial: Laparotomy (Active Comparator): Under general anesthesia in the NICU or operating room, a laparotomy will be performed following standard procedures.
  Interventions: Procedure: Laparotomy
- Randomized Trial: Peritoneal drain placement (Active Comparator): Place a one-fourth inch Penrose drain in the lower abdomen with local anesthesia and sedation.
  Interventions: Procedure: Drainage
- Preference Cohort: Laparotomy (Active Comparator): Under general anesthesia in the NICU or operating room, a laparotomy will be performed following standard procedures.
  Interventions: Procedure: Laparotomy
- Preference Cohort: Peritoneal drain placement (Active Comparator): Place a one-fourth inch Penrose drain in the lower abdomen with local anesthesia and sedation.
  Interventions: Procedure: Drainage

INTERVENTIONS:
Procedure: Laparotomy — Initial laparotomy will be performed. Standard procedures will be used, including inspection of the bowel with removal of diseased areas, creation of stoma(s), and other procedures deemed indicated by the surgeon.
  Arms: Preference Cohort: Laparotomy; Randomized Trial: Laparotomy
Procedure: Drainage — Initial drainage will involve placing a Penrose drain in the abdomen.
  Other Names: Peritoneal drain
  Arms: Preference Cohort: Peritoneal drain placement; Randomized Trial: Peritoneal drain placement

SUMMARY:
This study will compare the effectiveness of two surgical procedures -laparotomy versus drainage - commonly used to treat necrotizing enterocolitis (NEC) or isolated intestinal perforations (IP) in extremely low birth weight infants (≤1,000 g). Infants diagnosed with NEC or IP requiring surgical intervention, will be recruited. Subjects will be randomized to receive either a laparotomy or peritoneal drainage. Primary outcome is impairment-free survival at 18-22 months corrected age.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is a condition, generally affecting premature infants, in which the intestines become ischemic (lack oxygen and/or blood flow). NEC occurs in up to 5-15% of extremely low birth weight (ELBW) infants. Isolated or focal intestinal perforation (IP) is a less common condition, affecting an estimated 4% of ELBWs, in which a hole develops in the intestines leaking fluid into the abdominal cavity. Outcome for infants with NEC and/or IP is poor: 49% die and half of the surviving infants are neurodevelopmentally impaired.

Surgical options for NEC and IP include two possible procedures: peritoneal drainage, in which a tube is placed in the abdominal cavity through a small incision for fluid to drain out; or laparotomy, in which an incision is made in the abdomen and necrotic intestine is removed. Drainage may be followed by a laparotomy.

The Neonatal Research Network's observational study of 156 ELBW infants with NEC or IP (Pediatrics. 2006 Apr; 117(4): e680-7) showed comparable outcomes for the two procedures before hospital discharge, but suggested an advantage of laparotomy over drainage at 18-22 months corrected age with lower rates of death or neurodevelopmental impairment. However, the infants that underwent laparotomy were more mature; infants with drains were smaller and more premature. We hypothesize that initial laparotomy may improve an infant's long-term neurodevelopmental outcome, potentially by reducing the maximum severity or duration of inflammation.

This study included a randomized controlled trial to compare the effectiveness of laparotomy versus drainage for treating NEC or IP in extremely low birth weight infants. Target enrollment is 300 infants diagnosed with NEC or IP for randomization to receive initially either a laparotomy or drainage. Subsequent laparotomies may be performed on infants in either group, if their condition continues to deteriorate. Surviving infants will return for a follow-up assessment at 18-22 months corrected age.

This study also attempted to use a comprehensive cohort design that would have added additional information beyond the conventional randomized trial component. The cohort component included trial data among eligible, non-randomized infants with NEC/IP, who consented for the non-randomized cohort, would be collected and analyzed as a secondary specific aim. This additional cohort was called the preference cohort.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at ≤1,000 g birth weight
* Infant is ≤8 0/7 weeks of age at the time of eligibility assessment
* Pediatric surgeon decision to perform surgery for suspected NEC or IP
* Subject is at a center able to perform both laparotomy and drainage

Exclusion Criteria:

* Major anomaly that influences likelihood of developing primary outcome or affects surgical treatment considerations
* Congenital infection
* Prior laparotomy or peritoneal drain placement
* Prior NEC or IP
* Infant for whom full support is not being provided
* Follow-up unlikely

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 529 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; C. Michael Cotten, MD, Principal Investigator — Duke University; David Carlton, MD, Principal Investigator — Emory University; Greg Sokol, MD, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Frantz III, MD, Principal Investigator — Tufts Medical Center; Brenda Poindexter, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Bell, MD, Principal Investigator — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Myra Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Martin K. Blakely, MD, Study Director — Vanderbilt University Medical Center; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Barbara Schmidt, MD, MSc, Principal Investigator — Univeristy of Pennsylvania; Carl D'Angio, MD, Principal Investigator — University of Rochester; Uday Devaskar, MD, Principal Investigator — University of Carlifornia - Los Angeles; Leif Nelin, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; Brad Yoder, MD, Principal Investigator — University of Utah
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Rysavy MA, Eggleston B, Dahabreh IJ, Tyson JE, Patel RM, Watterberg KL, Greenberg RG, Pedroza C, Trotta M, Stevenson DK, Stoll BJ, Lally KP, Das A, Blakely ML; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Generalizability of the Necrotizing Enterocolitis Surgery Trial to the Target Population of Eligible Infants. J Pediatr. 2023 Nov;262:113453. doi: 10.1016/j.jpeds.2023.113453. Epub 2023 May 9. PMID 37169336
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Trial: Initial Laparotomy; Preference Cohort: Initial Laparotomy: Under general anesthesia in the neonatal intensive care unit (NICU) or operating room, a laparotomy will be performed following standard procedures.
- Randomized Trial: Initial Peritoneal Drain; Preference Cohort: Initial Peritoneal Drain: Place a one-fourth inch Penrose drain in the lower abdomen with local anesthesia and sedation.
Period: Overall Study
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain | Preference Cohort: Initial Laparotomy | Preference Cohort: Initial Peritoneal Drain
Started (Five infants in the preference cohort never received a Lap or Drain. These five infants are excluded from the summarization and analysis of preference cohort data.) | 148 | 162 | 100 | 119
Included in ITT Analysis | 146 | 162 | 100 | 119
Reached Network Status | 146 | 162 | 100 | 119
Completed (Primary Outcome Observed) | 141 | 154 | 93 | 115
Not Completed | 7 | 8 | 7 | 4
Not completed — Lost to Follow-up | 4 | 5 | 5 | 4
Not completed — Consent Withdrawn | 2 | 0 | 0 | 0
Not completed — Primary Outcome Indeterminate | 1 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Trial: Initial Laparotomy; Preference Cohort: Initial Laparotomy: Under general anesthesia in the NICU or operating room, a laparotomy will be performed following standard procedures.
- Total: Total of all reporting groups
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain | Preference Cohort: Initial Laparotomy | Preference Cohort: Initial Peritoneal Drain | Total
Number analyzed (Participants) | 146 | 162 | 100 | 119 | 527
Age, Continuous [Mean (Standard Deviation); unit: days] — Infant age at enrollment.
  days | 11.6 (10) | 12.1 (9.9) | 79.9 (125.4) | 49.9 (111.7) | 33.3 (81.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 66 | 63 | 48 | 53 | 230
  Male | 80 | 98 | 52 | 66 | 296
  Missing | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Maternal race because infant race not recorded
  Participants
    Black | 62 | 67 | 31 | 42 | 202
    Missing | 5 | 5 | 1 | 1 | 12
    Other | 6 | 8 | 9 | 6 | 29
    White | 73 | 82 | 59 | 70 | 284
Maternal hispanic ethnicity [Count of Participants; unit: Participants]
  Missing | 1 | 9 | 3 | 9 | 22
  No | 107 | 120 | 75 | 95 | 397
  Yes | 38 | 33 | 22 | 15 | 108
Infant gestational age [Mean (Standard Deviation); unit: weeks] | 25 (1.7) | 24.9 (1.7) | 24.6 (1.1) | 24.5 (1.2) | 25 (1.7)
Infant birth weight [Mean (Standard Deviation); unit: gram] | 721.2 (138.4) | 711.4 (135.9) | 719.8 (150.5) | 675.6 (161.7) | 707.6 (146.2)
Infant was small for gestational age [Count of Participants; unit: Participants]
  Missing | 0 | 1 | 0 | 0 | 1
  No | 131 | 145 | 84 | 98 | 458
  Yes | 15 | 16 | 16 | 21 | 68
Inborn status [Count of Participants; unit: Participants] — infant are inborn if they are born within the walls of one of the designated Neonatal Research Network (NRN) Network hospitals. An outborn infant is born at any other hospital, home delivery, taxi, etc.
  Participants
    In born | 82 | 90 | 65 | 75 | 312
    Out born | 64 | 72 | 35 | 44 | 215
Infant Apgar score at 1 minute [Median (Full Range); unit: units on a scale] — Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration" and scores range from 1 (worst) to 10 (best) indicating a baby's condition 1 minute after birth.
  units on a scale | 3 [0 to 9] | 3 [0 to 9] | 4 [2 to 6] | 4 [2 to 5] | 3 [0 to 9]
Infant Apgar score at 5 minute [Median (Full Range); unit: units on a scale] — Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration" and scores range from 1 (worst) to 10 (best) indicating a baby's condition 5 minutes after birth.
  units on a scale | 6 [0 to 9] | 6 [1 to 10] | 7 [5 to 8] | 7 [5 to 8] | 7 [0 to 10]
Infant had patent ductus arteriosus (PDA) prior to enrollment [Count of Participants; unit: Participants]
  Missing | 10 | 15 | 2 | 4 | 31
  No | 77 | 85 | 52 | 56 | 270
  Yes | 59 | 62 | 46 | 59 | 226
Infant received postnatal steroids [Count of Participants; unit: Participants]
  No | 119 | 115 | 67 | 83 | 384
  Yes | 27 | 47 | 33 | 36 | 143
Infant received indomethacin before or on Randomization [Count of Participants; unit: Participants]
  Missing | 3 | 6 | 3 | 7 | 19
  No | 69 | 74 | 51 | 38 | 232
  Yes | 74 | 82 | 46 | 74 | 276
Infant received enteral feedings before or on enrollment [Count of Participants; unit: Participants]
  Missing | 33 | 38 | 16 | 25 | 112
  No | 23 | 29 | 5 | 11 | 68
  Yes | 90 | 95 | 79 | 83 | 347
Infant had early onset sepsis before or on enrollment [Count of Participants; unit: Participants]
  Missing | 2 | 5 | 0 | 1 | 8
  No | 143 | 151 | 98 | 117 | 509
  Yes | 1 | 6 | 2 | 1 | 10
Infant had late onset sepsis before or on enrollment [Count of Participants; unit: Participants]
  Missing | 0 | 2 | 1 | 0 | 3
  No | 109 | 113 | 72 | 76 | 370
  Yes | 37 | 47 | 27 | 43 | 154
Infant had severe intraventricular hemorrhage (IVH) (grade 3 or 4) [Count of Participants; unit: Participants] — Severe IVH is defined as IVH Grades 3 or 4 on either side of the brain. The evaluation for IVH occurs early (within 28 days from birth) via a cranial sonogram and is classified as described by Papile.
  Participants
    Missing | 6 | 5 | 1 | 4 | 16
    No | 123 | 134 | 86 | 88 | 431
    Yes | 17 | 23 | 13 | 27 | 80
Infant on vasopressors at Enrollment [Count of Participants; unit: Participants]
  No | 105 | 103 | 55 | 71 | 334
  Yes | 41 | 59 | 45 | 47 | 192
  Missing | 0 | 0 | 0 | 1 | 1
Infant received HFOV or HFJV at randomization [Count of Participants; unit: Participants] — HFOV: high frequency oscillatory ventilation. HFJV: high frequency jet ventilation.
  Participants
    No | 114 | 114 | 51 | 66 | 345
    Yes | 32 | 48 | 49 | 53 | 182
Infant pH closest to enrollment [Mean (Standard Deviation); unit: pH] | 7.2 (0.1) | 7.2 (0.1) | 7.2 (0.1) | 7.2 (0.2) | 7.2 (0.1)
Infant fraction of inspired oxygen (FiO2) closest to enrollment [Mean (Standard Deviation); unit: Percent] | 44.8 (26.3) | 45.9 (24.1) | 57.8 (29.7) | 53.5 (30.0) | 49.6 (27.6)
Infant mean blood pressure [Mean (Standard Deviation); unit: mmHG] — The mean arterial blood pressure closest to the time of surgical consultation.
  mmHG | 37.1 (10.3) | 37.0 (11.5) | 39.0 (11.3) | 36.1 (11.7) | 37.2 (11.2)
Infant lowest platelet count [Mean (Standard Deviation); unit: 1000 platelets per microliter] | 155.7 (96) | 150.4 (80.9) | 156.2 (91.4) | 131.5 (79.6) | 148.7 (87.3)
Infant baseline risk of death or neurodevelopmental impairment (NDI) [Median (Standard Deviation); unit: Percent probability] — Infants randomized into NEST were stratified on a predicted probability of death or NDI. This predicted probability was based on a logistic regression model including birth weight, gestational age, vasopressor (yes/no), HFOV/HFJV (yes/no), pH, FiO2, and pre-operative diagnosis (NEC or IP). The predicted probability of death or NDI given these baseline measures is summarized in this variable.
  Percent probability | 63.4 (27) | 70.7 (23.7) | 88.1 (20.7) | 85.8 (23.1) | 70.3 (25.0)
Infant preoperative diagnosis (NEC or IP) [Count of Participants; unit: Participants] — Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP)
  Participants
    IP | 104 | 109 | 25 | 72 | 310
    NEC | 42 | 53 | 75 | 47 | 217
Maternal Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (6.7) | 27.3 (6.3) | 26.7 (6.3) | 26.8 (6.2) | 27.2 (6.4)
Married, Customized [Count of Participants; unit: Participants]
  Missing | 1 | 6 | 4 | 4 | 15
  No | 81 | 95 | 50 | 62 | 288
  Yes | 64 | 61 | 46 | 53 | 224
Maternal Education, Customized [Count of Participants; unit: Participants]
  College graduate | 18 | 21 | 19 | 25 | 83
  High school graduate | 42 | 38 | 19 | 25 | 124
  Less than high school | 21 | 28 | 22 | 12 | 83
  Missing | 42 | 51 | 25 | 38 | 156
  Some college | 23 | 24 | 15 | 19 | 81
Mother had private insurance [Count of Participants; unit: Participants]
  Missing | 0 | 3 | 0 | 1 | 4
  No | 98 | 113 | 71 | 65 | 347
  Yes | 48 | 46 | 29 | 53 | 176
Mother received prenatal care [Count of Participants; unit: Participants]
  Missing | 1 | 3 | 6 | 5 | 15
  No | 3 | 10 | 2 | 5 | 20
  Yes | 142 | 149 | 92 | 109 | 492
Mother received antibiotics [Count of Participants; unit: Participants]
  Missing | 28 | 37 | 15 | 18 | 98
  No | 39 | 42 | 19 | 19 | 119
  Yes | 79 | 83 | 66 | 82 | 310
Rupture of membranes > 18 hours [Count of Participants; unit: Participants]
  Missing | 22 | 29 | 7 | 6 | 64
  No | 101 | 108 | 69 | 97 | 375
  Yes | 23 | 25 | 24 | 16 | 88
Maternal hypertension [Count of Participants; unit: Participants]
  Missing | 26 | 31 | 10 | 13 | 80
  No | 85 | 98 | 65 | 84 | 332
  Yes | 35 | 33 | 25 | 22 | 115
Mother received antenatal magnesium [Count of Participants; unit: Participants]
  Missing | 52 | 68 | 59 | 66 | 245
  No | 17 | 21 | 6 | 7 | 51
  Yes | 77 | 73 | 35 | 46 | 231
Mother received steroids [Count of Participants; unit: Participants]
  Missing | 0 | 1 | 0 | 0 | 1
  No | 22 | 31 | 11 | 18 | 82
  Yes | 124 | 130 | 89 | 101 | 444

OUTCOME MEASURES:

1. Primary Outcome: Death or Neurodevelopmental Impairment (NDI)
Description: Death or NDI at 18-22 months corrected age
Time Frame: at 18-22 months corrected age
Population: Analysis of randomized trial data included all eligible participants who were consented, randomized, did not withdraw consent, and who provided outcome data after randomization. Analysis of preference cohort data included all eligible participants who were consented, enrolled, did not withdraw consent, and who provided outcome data.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain | Preference Cohort: Laparotomy | Preference Cohort: Initial Peritoneal Drain
Number analyzed (Participants) | 141 | 154 | 93 | 115
Participants
  No | 44 | 46 | 27 | 28
  Yes | 97 | 108 | 66 | 87
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis. Model included treatment, baseline risk of death or NDI, and pre-operative diagnosis (Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP)) as covariates; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.87 to 1.14] — RR: Initial Laparotomy over Peritoneal Drain. RR from robust Poisson regression with log link, reference cell coding, center as repeated measure. Model included treatment, baseline risk of death or NDI, and pre-op diagnosis (NEC/IP) as covariates
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis. Using Robust Poisson regression with log link and center as repeated measure, and effect coding, test for an interaction between treatment (Initial Laparotomy/Initial Peritoneal Drain) and pre-operative diagnosis (Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP)) as covariates. Model included treatment, baseline risk of death or NDI, pre-op diagnosis (NEC/IP), and treatment by pre-operative diagnosis as covariates; Test type: Other; p = 0.03, Robust Poisson regression — Pre-specified threshold = 0.05
Statistical Analysis 3: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A Bayesian analysis. Initial Laparotomy and Initial Peritoneal Drain were compared using log-binomial regression. The SAS procedure PROC MCMC with reference cell coding was used. Center (random effect), treatment, pre-operative diagnosis, and baseline risk of death or NDI were binary covariates. Pre-operative diagnosis levels were NEC and IP. Markov chain Monte Carlo (MCMC) characteristics: three chains, 10000 tunings, 10000 burn-ins, 1000000 samples, thinning=20; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.95, 95% credible interval of (0.82, 1.11)
Statistical Analysis 4: Comparison: Preference Cohort: Laparotomy vs Preference Cohort: Initial Peritoneal Drain; A frequentist analysis. Model included treatment, baseline risk of death or NDI, and pre-operative diagnosis (Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP)) covariates; Test type: Superiority; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.75 to 1.26] — RR: Initial Laparotomy over Peritoneal Drain. RR from robust regression with log link, reference cell coding, center as repeated measure. Model included treatment, baseline risk of death or NDI, and pre-op diagnosis (NEC/IP) as covariate

2. Secondary Outcome: Death
Description: Death by 18-22 months corrected age
Time Frame: by 18-22 months corrected age
Population: Analysis included all eligible participants who were consented, randomized, did not withdraw consent, and who provided outcome data after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  No | 105 | 114
  Yes | 41 | 48
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.69 to 1.45] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; Test type: Superiority — A Bayesian analysis. Initial Laparotomy and Initial Peritoneal Drain were compared using log-binomial regression. The SAS procedure PROC MCMC with reference cell coding was used. Center (random effect), treatment, pre-operative diagnosis, and baseline risk of death or NDI were binary covariates. Pre-operative diagnosis levels were NEC and IP. Markov chain Monte Carlo (MCMC) characteristics: three chains, 10000 tunings, 10000 burn-ins, 1000000 samples, thinning=20; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.95, 95% credible interval of (0.69, 1.30)

3. Secondary Outcome: Survival With Neurodevelopmental Impairment (NDI)
Description: NDI at 18-22 months corrected age (among survivors)
Time Frame: by 18-22 months corrected age
Population: Analysis included all eligible participants who were consented, randomized, did not withdraw consent, survived until follow-up visit at 18-22 months, and provided sufficient information to determine if NDI occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 100 | 106
Participants
  No | 44 | 46
  Yes | 56 | 60
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis. Estimate based on model fit using only data from study survivors; Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.78 to 1.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A Bayesian analysis among study survivors. Initial Laparotomy and Initial Peritoneal Drain were compared using log-binomial regression. The SAS procedure PROC MCMC with reference cell coding was used. Center (random effect), treatment, pre-operative diagnosis, and baseline risk of death or NDI were binary covariates. Pre-operative diagnosis levels were NEC and IP. Markov chain Monte Carlo (MCMC) characteristics: three chains, 10000 tunings, 10000 burn-ins, 1000000 samples, thinning=20; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.99, 95% credible interval of (0.78, 1.25)

4. Secondary Outcome: Death or Moderate to Severe Cerebral Palsy
Description: Death within 18-22 months corrected age or moderate to severe cerebral palsy at 18-22 months corrected age
Time Frame: up to the follow-up visit completed within the 18-22 months corrected age window
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 142 | 157
Participants
  No | 84 | 78
  Yes | 58 | 79
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.66 to 1.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.82, 95% credible interval of (0.65, 1.02)

5. Secondary Outcome: Death or Bayley Cognitive Composite Score Less Than 85
Description: Death within 18-22 months corrected age or Bayley cognitive composite score less than 85 at 18-22 months corrected age. Higher values of the Bayley cognitive composite score is better than lower values. Normal values are greater than or equal to 85. A moderate value is in the 70-84 range, and a severe value is <70.
Time Frame: up to the follow-up visit completed within the 18-22 months corrected age window
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 141 | 151
Participants
  No | 46 | 51
  Yes | 95 | 100
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.89 to 1.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.98, 95% credible interval of (0.84, 1.15)

6. Secondary Outcome: Death or Blindness
Description: Death within 18-22 months corrected age or blindness at 18-22 months corrected age
Time Frame: up to the follow-up visit completed within the 18-22 months corrected age window
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 142 | 157
Participants
  No | 101 | 105
  Yes | 41 | 52
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.64 to 1.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.86, 95% credible interval of (0.64, 1.16)

7. Secondary Outcome: Death or Hearing Loss
Description: Death within 18-22 months corrected age or hearing loss at 18-22 months corrected age
Time Frame: up to the follow-up visit completed within the 18-22 months corrected age window
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 141 | 156
Participants
  No | 98 | 105
  Yes | 43 | 51
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.69 to 1.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.92, 95% credible interval of (0.68, 1.25)

8. Secondary Outcome: Subsequent Laparotomy
Description: Subsequent laparotomy after initial surgery
Time Frame: between initial surgery and Neonatal Research Network NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 145 | 162
Participants
  No | 110 | 81
  Yes | 35 | 81
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 0.47, 95% CI 2-sided [0.35 to 0.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.51, 95% credible interval of (0.37, 0.69)

9. Secondary Outcome: Any Intraoperative Complications During Any Surgery
Description: Any intraoperative complications during any surgery
Time Frame: between randomization and Neonatal Research Network NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 145 | 162
Participants
  No | 116 | 141
  Yes | 29 | 21
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 1.57, 95% CI 2-sided [1.04 to 2.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.45, 95% credible interval of (0.92, 2.31)

10. Secondary Outcome: Any Wound Dehiscence
Description: Any wound dehiscence during any surgery
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  No | 135 | 154
  Yes | 11 | 8
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 1.58, 95% CI 2-sided [0.71 to 3.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.31, 95% credible interval of (0.66, 2.62)

11. Secondary Outcome: Any Intra-abdominal Abscess
Description: Any intra-abdominal abscess during any surgery
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  No | 141 | 158
  Yes | 5 | 4
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; This analysis used model identical to other by treatment analyses for binary outcome. RR estimated from robust Poisson regression with log link, reference cell coding, center as repeated measure. RR: Initial Laparotomy over Peritoneal Drain. Model included treatment, baseline risk of death or NDI, and pre-op diagnosis (NEC/IP) as covariates. However, adjusted RR estimates could not be calculated due to the iteration limit being excessed in PROC GENMOD
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.16, 95% credible interval of (0.50, 2.65)

12. Secondary Outcome: Any Intestinal Stricture
Description: Any intestinal stricture during any surgery
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  No | 139 | 153
  Yes | 7 | 9
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.34 to 2.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.93, 95% credible interval of (0.45, 1.91)

13. Secondary Outcome: Any Late Onset Sepsis
Description: Any late onset sepsis after randomization
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 160
Participants
  No | 123 | 126
  Yes | 23 | 34
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.37 to 1.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.75, 95% credible interval of (0.48, 1.16)

14. Secondary Outcome: Any Parenteral Nutrition (PN)-Associated Cholestasis
Description: Any Parenteral nutrition (PN)-associated cholestasis during any surgery
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  No | 110 | 116
  Yes | 36 | 46
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.70 to 1.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A Bayesian analysis. Initial Laparotomy and Initial Peritoneal Drain were compared using log-binomial regression. The SAS procedure PROC MCMC with effect coding was used. Center (random effect), treatment, pre-operative diagnosis, and baseline risk of death or NDI were binary covariates. Pre-operative diagnosis levels were NEC and IP. Markov chain Monte Carlo (MCMC) characteristics: three chains, 10000 tunings, 10000 burn-ins, 1000000 samples, thinning=20; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.91, 95% credible interval of (0.65, 1.27)

15. Secondary Outcome: Any Severe IVH
Description: Any severe IVH ater randomization
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 140 | 157
Participants
  No | 122 | 132
  Yes | 18 | 25
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.44 to 1.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.82, 95% credible interval of (0.49, 1.33)

16. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration of mechanical ventilation while on study
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 107 | 120
days | 33.3 (25.6) | 38.9 (26.7)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Mean Difference (Final Values) = -6.01, 95% CI 2-sided [-12.77 to 0.75] — Mean Difference (MD): Laparotomy minus Drain. MD from mixed model using PROC MIXED in SAS, center as random effect, and reference cell coding. Model included treatment, baseline risk of death or NDI, and pre-op diagnosis (NEC/IP) as covariates
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A Bayesian analysis. Initial Laparotomy and Initial Peritoneal Drain were compared using a hierarchical linear regression. The SAS procedure PROC MCMC with reference cell coding was used. Center (random effect), treatment, pre-operative diagnosis, and baseline risk of death or NDI were binary covariates. Pre-operative diagnosis levels were NEC and IP. Markov chain Monte Carlo (MCMC) characteristics: three chains, 10000 tunings, 10000 burn-ins, 1000000 samples, thinning=20; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=1000), treatment, baseline risk, and preop diagnosis parameters = Normal(mean=0, variance=10), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median difference Initial Laparotomy minus Initial Drainage was -2.68, 95% credible interval of (-7.11, 1.83)

17. Secondary Outcome: Duration of Parenteral Nutrition
Description: Duration of parenteral nutrition while on study
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 135 | 149
days | 55.5 (34.1) | 64.1 (36.4)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Mean Difference (Final Values) = -8.75, 95% CI 2-sided [-17.05 to -0.46] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 16, analysis 2]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=1000), treatment, baseline risk, and preop diagnosis parameters = Normal(mean=0, variance=10), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median difference Initial Laparotomy minus Initial Drainage was -3.23, 95% credible interval of (-8.08, 1.68)

18. Secondary Outcome: Final Bowel Length
Description: Final bowel length after last surgery
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 28 | 16
cm | 74.4 (24.6) | 68.7 (35.7)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Mean Difference (Final Values) = 6.59, 95% CI 2-sided [-9.09 to 22.27] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A Bayesian analysis. Initial Laparotomy and Initial Peritoneal Drain were compared using a hierarchical linear regression. The SAS procedure PROC MCMC with reference coding was used. Center (random effect), treatment, pre-operative diagnosis, and baseline risk of death or NDI were binary covariates. Pre-operative diagnosis levels were NEC and IP. Markov chain Monte Carlo (MCMC) characteristics: three chains, 10000 tunings, 10000 burn-ins, 1000000 samples, thinning=20; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=1000), treatment, baseline risk, and preop diagnosis parameters = Normal(mean=0, variance=10), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median difference Initial Laparotomy minus Initial Drainage was 1.65, 95% credible interval of (-3.97, 7.23)

19. Secondary Outcome: Time to Full Feeds
Description: Time to full feeds while on study
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 92 | 92
days | 46.9 (45.8) | 50.6 (27.7)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-13.02 to 7.91] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 16, analysis 2]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=1000), treatment, baseline risk, and preop diagnosis parameters = Normal(mean=0, variance=10), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median difference Initial Laparotomy minus Initial Drainage was -0.71, 95% credible interval of (-5.89, 4.48)

20. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay while on study
Time Frame: from randomization up to 1 year following birth
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 137 | 156
days | 101.2 (71.2) | 113.8 (73.8)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A frequentist analysis; Test type: Superiority; Mean Difference (Final Values) = -13.95, 95% CI 2-sided [-30.54 to 2.63] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 16, analysis 2]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=1000), treatment, baseline risk, and preop diagnosis parameters = Normal(mean=0, variance=10), random effect standard deviation = Half-Normal(mean=0, variance=10). The posterior median difference Initial Laparotomy minus Initial Drainage was -1.78, 95% credible interval of (-7.44, 3.87)

21. Secondary Outcome: Death or NDI Stratified by Pre-operative Diagnosis
Description: Death or NDI at 18-22 months corrected age. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: at 18-22 months corrected age
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 141 | 154
Participants
  IP: number analyzed (Participants) | 99 | 102
  IP: No | 31 | 38
  IP: Yes | 68 | 64
  NEC: number analyzed (Participants) | 42 | 52
  NEC: No | 13 | 8
  NEC: Yes | 29 | 44
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; This by treatment and by pre-operative diagnosis secondary analysis was completed by using a robust Poisson regression model, with log link and center as repeated measure. Model included treatment, baseline risk of death or NDI, pre-op diagnosis (NEC/IP), and treatment by pre-op diagnosis as covariates. Reported results in this analysis restricted to model based treatment effect estimate (laparotomy over drain) when pre-operative diagnosis is equal to NEC; Test type: Superiority; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.64 to 1.04] — The model was fit using PROC GENMOD in SAS, using center as the repeated effect. Effect coding was used to represent the binary covariates
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; This by treatment and by pre-operative diagnosis secondary analysis was completed by using a robust Poisson regression model, with log link and center as repeated measure. Model included treatment, baseline risk of death or NDI, pre-op diagnosis (NEC/IP), and treatment by pre-op diagnosis as covariates. Reported results in this analysis restricted to model based treatment effect estimate (laparotomy over drain) when pre-operative diagnosis is equal to IP; Test type: Superiority; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.95 to 1.31] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A Bayesian analysis. Within pre-operative diagnosis, Initial Laparotomy and Initial Peritoneal Drain were compared using log-binomial regression. Pre-operative diagnosis levels were NEC and IP. PROC MCMC with effect coding was used. Center (random effect), treatment, pre-operative diagnosis, baseline risk, and the treatment by Preoperative diagnosis were the covariates. Markov chain Monte Carlo (MCMC) characteristics: three chains, 10000 tunings, 10000 burn-ins, 1000000 samples, thinning=20; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). For the NEC pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.81, 95% credible interval of (0.63, 1.00). For the IP pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.09, 95% credible interval of (0.90, 1.33)

22. Secondary Outcome: Death Stratified by Pre-operative Diagnosis
Description: Death within 18-22 months corrected age. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: by 18-22 months corrected age
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  IP: number analyzed (Participants) | 104 | 109
  IP: No | 80 | 88
  IP: Yes | 24 | 21
  NEC: number analyzed (Participants) | 42 | 53
  NEC: No | 25 | 26
  NEC: Yes | 17 | 27
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.52 to 1.13] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.28, 95% CI 2-sided [0.79 to 2.06] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). For the NEC pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.82, 95% credible interval of (0.53, 1.20). For the IP pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.18, 95% credible interval of (0.74, 1.87)

23. Secondary Outcome: Survival With Neurodevelopmental Impairment (NDI) Stratified by Pre-operative Diagnosis
Description: NDI at 18-22 months corrected age (among survivors). Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: by 18-22 months corrected age
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 100 | 106
Participants
  IP: number analyzed (Participants) | 75 | 81
  IP: No | 31 | 38
  IP: Yes | 44 | 43
  NEC: number analyzed (Participants) | 25 | 25
  NEC: No | 13 | 8
  NEC: Yes | 12 | 17
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.42 to 1.27] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.85 to 1.45] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; A Bayesian analysis. Within pre-operative diagnosis, Initial Laparotomy and Initial Peritoneal Drain were compared using log-binomial regression. Pre-operative diagnosis levels were NEC and IP. PROC MCMC with effect coding was used. Center (random effect), treatment, pre-operative diagnosis, baseline risk, and the treatment by Pre-operative diagnosis were the covariates. Markov chain Monte Carlo (MCMC) characteristics: three chains, 10000 tunings, 10000 burn-ins, 1000000 samples, thinning=20; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). For the NEC pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.76, 95% credible interval of (0.48, 1.18). For the IP pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.08, 95% credible interval of (0.83, 1.42)

24. Secondary Outcome: Death or Moderate to Severe Cerebral Palsy Stratified by Pre-operative Diagnosis
Description: Death within 18-22 months corrected age or moderate to severe cerebral palsy at 18-22 months corrected age. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: up to the follow-up visit completed within the 18-22 months corrected age window
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 142 | 157
Participants
  IP: number analyzed (Participants) | 100 | 105
  IP: No | 64 | 64
  IP: Yes | 36 | 41
  NEC: number analyzed (Participants) | 42 | 52
  NEC: No | 20 | 14
  NEC: Yes | 22 | 38
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.47 to 1.05] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.76 to 1.19] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). For the NEC pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.73, 95% credible interval of (0.52, 0.96). For the IP pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.95, 95% credible interval of (0.68, 1.32)

25. Secondary Outcome: Death or Bayley Cognitive Composite Score Less Than 85 Stratified by Pre-operative Diagnosis
Description: Death within 18-22 months corrected age or Bayley cognitive composite score less than 85 at 18-22 months corrected age. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP). Higher values of the Bayley cognitive composite score is better than lower values. Normal values are greater than or equal to 85. A moderate value is in the 70-84 range, and a severe value is <70.
Time Frame: up to the follow-up visit completed within the 18-22 months corrected age window
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 141 | 151
Participants
  IP: number analyzed (Participants) | 99 | 101
  IP: No | 32 | 42
  IP: Yes | 67 | 59
  NEC: number analyzed (Participants) | 42 | 50
  NEC: No | 14 | 9
  NEC: Yes | 28 | 41
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.61 to 1.06] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.17, 95% CI 2-sided [1.01 to 1.37] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). For the NEC pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.80, 95% credible interval of (0.61, 1.01). For the IP pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.15, 95% credible interval of (0.94, 1.42)

26. Secondary Outcome: Death or Blindness Stratified by Pre-operative Diagnosis
Description: Death within 18-22 months corrected age or blindness at 18-22 months corrected age. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: up to the follow-up visit completed within the 18-22 months corrected age window
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 142 | 157
Participants
  IP: number analyzed (Participants) | 100 | 105
  IP: No | 76 | 83
  IP: Yes | 24 | 22
  NEC: number analyzed (Participants) | 42 | 52
  NEC: No | 25 | 22
  NEC: Yes | 17 | 30
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.46 to 1.01] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.22, 95% CI 2-sided [0.74 to 2.01] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). For the NEC pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.72, 95% credible interval of (0.48, 1.05). For the IP pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.12, 95% credible interval of (0.71, 1.76)

27. Secondary Outcome: Death or Hearing Loss Stratified by Pre-operative Diagnosis
Description: Death within 18-22 months corrected age or hearing loss at 18-22 months corrected age. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: up to the follow-up visit completed within the 18-22 months corrected age window
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 141 | 156
Participants
  IP: number analyzed (Participants) | 99 | 104
  IP: No | 73 | 81
  IP: Yes | 26 | 23
  NEC: number analyzed (Participants) | 42 | 52
  NEC: No | 25 | 24
  NEC: Yes | 17 | 28
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.51 to 1.04] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.25, 95% CI 2-sided [0.82 to 1.93] — The model was fit using PROC GENMOD in SAS, using center as the repeated effect. Effect coding was used to represent the binary covariates. Reported results in this analysis restricted to infants with IP
Statistical Analysis 3: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 3]; Test type: Superiority; Priors for model parameters: intercept = Normal(mean=0, variance=100), baseline risk and preop diagnosis parameters = Normal(mean=0, variance=1), treatment and the interaction term = Normal(mean=0, variance=0.31416), random effect standard deviation = Half-Normal(mean=0, variance=10). For the NEC pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 0.77, 95% credible interval of (0.51, 1.14). For the IP pre-operative diagnosis, the posterior median relative risk of Initial Laparotomy over Initial Drainage was 1.17, 95% credible interval of (0.76, 1.81)

28. Secondary Outcome: Subsequent Laparotomy Stratified by Pre-operative Diagnosis
Description: Subsequent laparotomy after initial surgery. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 145 | 162
Participants
  IP: number analyzed (Participants) | 104 | 109
  IP: No | 81 | 58
  IP: Yes | 23 | 51
  NEC: number analyzed (Participants) | 41 | 53
  NEC: No | 29 | 23
  NEC: Yes | 12 | 30
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.53, 95% CI 2-sided [0.31 to 0.89] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.44, 95% CI 2-sided [0.29 to 0.66] — [estimate comment as in outcome 21, analysis 1]

29. Secondary Outcome: Any Intraoperative Complications During Any Surgery Stratified by Pre-operative Diagnosis
Description: Any intraoperative complications during any surgery. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 145 | 162
Participants
  IP: number analyzed (Participants) | 104 | 109
  IP: No | 83 | 95
  IP: Yes | 21 | 14
  NEC: number analyzed (Participants) | 41 | 53
  NEC: No | 33 | 46
  NEC: Yes | 8 | 7
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.44, 95% CI 2-sided [0.58 to 3.57] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.63, 95% CI 2-sided [1.06 to 2.50] — [estimate comment as in outcome 21, analysis 1]

30. Secondary Outcome: Any Wound Dehiscence Stratified by Pre-operative Diagnosis
Description: Any wound dehiscence during any surgery. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  IP: number analyzed (Participants) | 104 | 109
  IP: No | 99 | 104
  IP: Yes | 5 | 5
  NEC: number analyzed (Participants) | 42 | 53
  NEC: No | 36 | 50
  NEC: Yes | 6 | 3
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 2.52, 95% CI 2-sided [0.84 to 7.55] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.38 to 2.88] — [estimate comment as in outcome 21, analysis 1]

31. Secondary Outcome: Any Intra-abdominal Abscess Stratified by Pre-operative Diagnosis
Description: Any intra-abdominal abscess during any surgery. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  IP: number analyzed (Participants) | 104 | 109
  IP: No | 101 | 106
  IP: Yes | 3 | 3
  NEC: number analyzed (Participants) | 42 | 53
  NEC: No | 40 | 52
  NEC: Yes | 2 | 1
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.78, 95% CI 2-sided [0.82 to 3.86] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.42 to 3.20] — [estimate comment as in outcome 21, analysis 1]

32. Secondary Outcome: Any Intestinal Stricture Stratified by Pre-operative Diagnosis
Description: Any intestinal stricture during any surgery. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  IP: number analyzed (Participants) | 104 | 109
  IP: No | 101 | 103
  IP: Yes | 3 | 6
  NEC: number analyzed (Participants) | 42 | 53
  NEC: No | 38 | 50
  NEC: Yes | 4 | 3
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.68, 95% CI 2-sided [0.35 to 8.05] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.10 to 2.44] — [estimate comment as in outcome 21, analysis 1]

33. Secondary Outcome: Any Late Onset Sepsis Stratified by Pre-operative Diagnosis
Description: Any late onset sepsis after randomization. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 160
Participants
  IP: number analyzed (Participants) | 104 | 107
  IP: No | 88 | 80
  IP: Yes | 16 | 27
  NEC: number analyzed (Participants) | 42 | 53
  NEC: No | 35 | 46
  NEC: Yes | 7 | 7
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.62 to 2.69] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.60, 95% CI 2-sided [0.27 to 1.32] — [estimate comment as in outcome 21, analysis 1]

34. Secondary Outcome: Any Parenteral Nutrition (PN)-Associated Cholestasis Stratified by Pre-operative Diagnosis
Description: Any Parenteral nutrition (PN)-associated cholestasis during any surgery. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 146 | 162
Participants
  IP: number analyzed (Participants) | 104 | 109
  IP: No | 79 | 82
  IP: Yes | 25 | 27
  NEC: number analyzed (Participants) | 42 | 53
  NEC: No | 31 | 34
  NEC: Yes | 11 | 19
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.41 to 1.36] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.69 to 1.42] — [estimate comment as in outcome 21, analysis 1]

35. Secondary Outcome: Any Severe IVH Stratified by Pre-operative Diagnosis
Description: Any severe IVH ater randomization. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 140 | 157
Participants
  IP: number analyzed (Participants) | 101 | 106
  IP: No | 84 | 84
  IP: Yes | 17 | 22
  NEC: number analyzed (Participants) | 39 | 51
  NEC: No | 38 | 48
  NEC: Yes | 1 | 3
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.43, 95% CI 2-sided [0.04 to 4.45] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 21, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.44 to 1.49] — [estimate comment as in outcome 21, analysis 1]

36. Secondary Outcome: Duration of Mechanical Ventilation Stratified by Pre-operative Diagnosis
Description: Duration of mechanical ventilation while on study. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 107 | 120
days
  IP: number analyzed (Participants) | 80 | 82
  IP | 34.1 (26.6) | 42.2 (28)
  NEC: number analyzed (Participants) | 27 | 38
  NEC | 31 (22.6) | 31.7 (22.5)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; This by treatment and by pre-operative diagnosis secondary analysis was completed by using a mixed linear regression model, using center as the random effect. Model included treatment, baseline risk of death or NDI, pre-op diagnosis (NEC/IP), and treatment by pre-op diagnosis as covariates. Reported results in this analysis restricted to model based treatment effect estimate (laparotomy minus drain) when pre-operative diagnosis is equal to NEC; Test type: Superiority; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-14.10 to 11.60] — The model was fit using PROC MIXED in SAS, using center as the random effect. Effect coding was used to represent the binary covariates
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; This by treatment and by pre-operative diagnosis secondary analysis was completed by using a mixed linear regression model, using center as the random effect. Model included treatment, baseline risk of death or NDI, pre-op diagnosis (NEC/IP), and treatment by pre-op diagnosis as covariates. Reported results in this analysis restricted to model based treatment effect estimate (laparotomy minus drain) when pre-operative diagnosis is equal to IP; Test type: Superiority; Mean Difference (Final Values) = -7.85, 95% CI 2-sided [-15.84 to 0.13] — [estimate comment as in outcome 36, analysis 1]

37. Secondary Outcome: Duration of Parenteral Nutrition Stratified by Pre-operative Diagnosis
Description: Duration of parenteral nutrition while on study. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 135 | 149
days
  IP: number analyzed (Participants) | 100 | 102
  IP | 56.3 (35.2) | 63.6 (33.7)
  NEC: number analyzed (Participants) | 35 | 47
  NEC | 53.5 (31.3) | 65.3 (42)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -11.57, 95% CI 2-sided [-27.15 to 4.01] — [estimate comment as in outcome 36, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 36, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -7.63, 95% CI 2-sided [-17.46 to 2.20] — [estimate comment as in outcome 36, analysis 1]

38. Secondary Outcome: Final Bowel Length Stratified by Pre-operative Diagnosis
Description: Final bowel length after last surgery. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 28 | 16
cm
  IP: number analyzed (Participants) | 16 | 7
  IP | 83.1 (20.9) | 74.7 (22.4)
  NEC: number analyzed (Participants) | 12 | 9
  NEC | 62.7 (25) | 64 (44.2)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 4.00, 95% CI 2-sided [-18.84 to 26.83] — [estimate comment as in outcome 36, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 36, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = 9.05, 95% CI 2-sided [-13.29 to 31.38] — [estimate comment as in outcome 36, analysis 1]

39. Secondary Outcome: Time to Full Feeds Stratified by Pre-operative Diagnosis
Description: Time to full feeds while on study. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 92 | 92
days
  IP: number analyzed (Participants) | 70 | 70
  IP | 52.4 (50.4) | 56.3 (27.1)
  NEC: number analyzed (Participants) | 22 | 22
  NEC | 29.6 (18.9) | 32.3 (21.3)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -3.13, 95% CI 2-sided [-24.62 to 18.36] — [estimate comment as in outcome 36, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 36, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -2.39, 95% CI 2-sided [-14.42 to 9.63] — The model was fit using PROC MIXED in SAS, using center as the random effect. Effect coding was used to represent the binary covariates. Reported results in this analysis restricted to infants with IP

40. Secondary Outcome: Length of Hospital Stay Stratified by Pre-operative Diagnosis
Description: Length of hospital stay while on study. Stratification variable is pre-operative diagnosis: Necrotizing Enterocolitis (NEC) or Isolated Intestinal Perforation (IP).
Time Frame: from randomization up to 1 year following birth
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain
Number analyzed (Participants) | 137 | 156
days
  IP: number analyzed (Participants) | 98 | 103
  IP | 109.6 (67) | 121.3 (64.7)
  NEC: number analyzed (Participants) | 39 | 53
  NEC | 80.2 (77.8) | 99.2 (87.7)
Statistical Analysis 1: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -18.43, 95% CI 2-sided [-48.41 to 11.55] — [estimate comment as in outcome 36, analysis 1]
Statistical Analysis 2: Comparison: Randomized Trial: Initial Laparotomy vs Randomized Trial: Initial Peritoneal Drain; [analysis description as in outcome 36, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -11.95, 95% CI 2-sided [-31.96 to 8.06] — [estimate comment as in outcome 36, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events are monitored from randomization through study status (death, discharge or 120 days)
Arm/Group | Randomized Trial: Initial Laparotomy | Randomized Trial: Initial Peritoneal Drain | Preference Cohort: Initial Laparotomy | Preference Cohort: Initial Peritoneal Drain
All-Cause Mortality (participants affected / at risk) | 41/146 | 48/162 | 48/100 | 60/119
Serious Adverse Events (participants affected / at risk) | 41/146 | 49/162 | 49/100 | 60/119
Other Adverse Events (participants affected / at risk) | 0/146 | 0/162 | 0/100 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Trial: Initial Laparotomy (N=146) | Randomized Trial: Initial Peritoneal Drain (N=162) | Preference Cohort: Initial Laparotomy (N=100) | Preference Cohort: Initial Peritoneal Drain (N=119)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal herniation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal spontaneous intestinal perforation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 9 (9)
Necrotizing enterocolitis neonatal (Gastrointestinal disorders) | 21 (21) | 24 (24) | 35 (35) | 25 (25)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
CNS injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal sepsis (Infections and infestations) | 10 (10) | 16 (16) | 13 (13) | 9 (9)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 7 (7)
Intracranial hemorrhage (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 3 (3)
Death (General disorders) | 4 (4) | 11 (11) | 6 (6) | 8 (8) — Babies who died but had no information about cause of death or an SEA record regarding the death was assigned SOC='General disorders' and PT='Death'
Fungal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prematurity (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Neonatal pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neonatal pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 7 (7)
Renal failure neonatal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiorgan failure (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coagulopathies (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication policies.

DOCUMENTS (3):
  • Study Protocol (2013-02-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT01029353/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT01029353/SAP_001.pdf
  • Informed Consent Form (2013-02-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT01029353/ICF_002.pdf